CLINICAL TRIAL: NCT02916888
Title: Patient and Caregiver Quality of Life in the Treatment of Atopic Dermatitis in Pediatric Patients: a Comparison Between a General Pediatric Practice and a Pediatric Dermatology Practice
Brief Title: A Study Comparing the Quality of Life of Patients in the Treatment of Eczema by Pediatric Generalists and Specialists
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1605017845
Record Dates: First submitted 2016-09-23; First posted 2016-09-28 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Eczema; Dermatitis; Dermatitis, Atopic; Genetic Disease, Inborn; Hypersensitivity; Hypersensitivity, Immediate; Immune System Diseases; Skin Diseases; Skin Diseases, Eczematous; Skin Diseases, Genetic
Keywords: Atopic dermatitis; Topical corticosteroid; Pediatric; Eczema; Quality of life
MeSH Terms: conditions — Eczema; Dermatitis; Dermatitis, Atopic; Genetic Diseases, Inborn; Hypersensitivity; Hypersensitivity, Immediate; Immune System Diseases; Skin Diseases; Skin Diseases, Eczematous; Skin Diseases, Genetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Saliva samples for salivary cortisol detection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Care provided by general pediatrician: Standard of care management of atopic dermatitis by general pediatrician. This includes an initial visit with a 2-week follow-up.
  Interventions: Other: Care provided by general pediatrician
- Care provided by pediatric dermatologist: Standard of care management of atopic dermatitis by pediatric dermatologist. This includes an initial visit with a 2-week follow-up.
  Interventions: Other: Care provided by pediatric dermatologist

INTERVENTIONS:
Other: Care provided by general pediatrician — Standard of care management of atopic dermatitis by a general pediatrician.
  Groups: Care provided by general pediatrician
Other: Care provided by pediatric dermatologist — Standard of care management of atopic dermatitis by a pediatric dermatologist.
  Groups: Care provided by pediatric dermatologist

SUMMARY:
The purpose of this study is to investigate the differences in the quality of life of patients and caregivers who are treated by general pediatricians versus pediatric dermatologists for eczema (atopic dermatitis or AD).

DETAILED DESCRIPTION:
Hypothesis:

We hypothesize that on average, the patients treated by the general pediatrician will have a smaller increase in quality of life at the end of the 2-week treatment period when compared to patients treated by the specialist.

Methods:

The primary endpoint will be the difference in patient and caregiver quality of life from baseline for the group treated by the general pediatrician and the group treated by the pediatric dermatologist. Secondary endpoints will be the difference in atopic dermatitis severity and TCS phobia from baseline.

Patients will be recruited from the Yale Pediatric Dermatology Clinic and Long Wharf Pediatrics and Adolescent Medicine in New Haven, CT.

Data Collection:

Assessment of AD by the investigator (EASI) and the patient/caregiver (POEM) will be completed at baseline on Day 0 in the clinic. Quality life measures (CDLQI/IDQoL/DFI) and steroid phobia measure (TOPICOP) will also be completed on Day 0. Follow-up clinical assessment will include skin examinations, and will be performed on Day 14. On the follow-up visit, the investigator will perform an assessment of AD severity using the EASI scoring method, ask patients/caregivers to re-take the CDLQI or IDQoL, DFI, POEM and TOPICOP, ask patients/caregivers to report adverse effects, and take digital photography utilizing the same standard poses as baseline. Patients' medication will be weighed to estimate amount of medication used in the 2-week treatment period. We will also instruct the patients and families to treat any subsequent AD flares in a similar manner as the first two weeks of the study, however they will treat until clear and may discontinue prior to 2 weeks of therapy.

Blinding:

This will be a single-blinded study. Patients will only know that there are 2 patient groups that are being treated by physicians, and that these 2 groups are being compared, but will not know that one group is being treated by a generalist and the other by a specialist. Given the study design, it will be impossible to blind investigators.

Treatment Administration:

There will be no research treatment/procedures that are not standard of care treatment. Standard of care treatment will be administered on an outpatient basis. All patients treated will receive a one-page handout, which briefly explains AD and educates families on how to prevent further atopic dermatitis outbreaks. All patients will also receive a page explaining how to apply corticosteroid ointment for treatment of AD.

Patients will adhere to twice daily administration of corticosteroid ointment for 2 weeks, and then will be assessed for clearance of AD. Caregivers or patients will document adherence at home daily in a chart that will be provided to them at their initial visit.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the clinical criteria for the diagnosis of atopic dermatitis
2. Have disease over at least 5% of their total body surface area.
3. Less than 7 years of age.
4. Families able to comprehend written instructions in English and able to complete questionnaires with assistance if needed.
5. Parents/guardians able to understand and willing to sign a parental permission form.

Exclusion Criteria:

1. Clinically infected atopic dermatitis.
2. Lack of follow-up after initial visit or regimen non-adherence.
3. Patients who are allergic or intolerant of the topical medications employed in this study.

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients under 7 years old that have atopic dermatitis from the Greater New Haven area.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in quality of life of patients | 2 weeks
  Measured using Infant's Dermatitis Quality of Life Index (IDQoL) or Children's Dermatology Life Quality Index(CDLQI) depending on age

SECONDARY OUTCOMES:
Change in quality of life of patient caregivers | 2 weeks
  Measured using Dermatitis Family Impact questionnaire (DFI)
Change in clinical severity of atopic dermatitis | 2 weeks
  Measured using Eczema Area and Severity Index (EASI) or Patient-Oriented Eczema Measure (POEM)
Change in topical corticosteroid phobia in caregivers | 2 weeks
  Measured using Topical Corticosteroid Phobia scale (TOPICOP)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Antaya, MD, Principal Investigator — Yale University
Locations (1):
- Yale Dermatology Associates, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eichenfield LF, Tom WL, Chamlin SL, Feldman SR, Hanifin JM, Simpson EL, Berger TG, Bergman JN, Cohen DE, Cooper KD, Cordoro KM, Davis DM, Krol A, Margolis DJ, Paller AS, Schwarzenberger K, Silverman RA, Williams HC, Elmets CA, Block J, Harrod CG, Smith Begolka W, Sidbury R. Guidelines of care for the management of atopic dermatitis: section 1. Diagnosis and assessment of atopic dermatitis. J Am Acad Dermatol. 2014 Feb;70(2):338-51. doi: 10.1016/j.jaad.2013.10.010. Epub 2013 Nov 27. PMID 24290431